CLINICAL TRIAL: NCT06572020
Title: The Effect of Simulation-Based Blood Pressure and Electrocardiography Training in Cardiac Rehabilitation on Physiotherapy Student's Self-Confidence and Satisfaction Level
Brief Title: The Effect of Simulation-Based Training on Physiotherapy Student's Self-Confidence and Satisfaction Level
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ACU-CASE-1
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Simulation of Physical Illness; Blood Pressure
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physiotherapy students (Experimental): Physiotherapy students
  Interventions: Other: education

INTERVENTIONS:
Other: education — simulation-based training on blood pressure and ECG measurement

SUMMARY:
The goal of this clinical trial is to investigate the effect of simulation-based training in the cardiac rehabilitation course on the confidence and satisfaction of physiotherapy and rehabilitation students.

The main questions it aims to answer are:

Does simulation-based training in blood pressure and electrocardiography in cardiac rehabilitation have an effect on the confidence levels of physiotherapy students? Does simulation-based training in blood pressure and electrocardiography in cardiac rehabilitation have an effect on the satisfaction levels of physiotherapy students? Does simulation-based training in blood pressure and electrocardiography in cardiac rehabilitation have an effect on the theoretical knowledge levels of physiotherapy students?

This study is planned to be conducted with 39 individuals who are enrolled in the course and taking it for the first time.

The study will be conducted at the Acıbadem University CASE Laboratory using surveys administered before and after simulation training on blood pressure and electrocardiography (ECG). The sociodemographic characteristics of the participants will be recorded using an information form. The level of experience, theoretical knowledge, and competency in blood pressure and ECG measurement will be assessed with a 'Pre-Test' prepared for this purpose. The same parameters, along with satisfaction with the simulation training, will be assessed with a 'Post-Test' using a self-assessment survey method after the training. The prepared surveys, detailed below, will be completed separately for blood pressure and ECG training.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of Physiotherapy and Rehabilitation at Acıbadem University
* Being enrolled in the Cardiac Diseases and Rehabilitation course
* Having completed the consent form

Exclusion Criteria:

* Repeating the Cardiac Diseases and Rehabilitation course
* Refusing to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-09-26 (Estimated)

PRIMARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning | One day (The assessments will be conducted once)
  The 'Student Satisfaction and Confidence Scale in Learning' will be administered separately for blood pressure and ECG training at the end of the simulation. The original 13-item scale by Jeffries and Rizzolo (2006) was adapted into Turkish with 12 items. It uses a 5-point Likert scale and includes two subscales: 'Satisfaction with Current Learning' (5 items) and 'Confidence in Learning' (7 items), with no negative items. Scores are obtained by averaging subscale scores. Higher total scores indicate greater satisfaction and confidence. Item 13 was recommended for exclusion by Franklin et al., re-evaluated by language experts, and removed by the research group. Therefore, the 12-item version will be used in our study

SECONDARY OUTCOMES:
Practitioner Competency Test | One day (The assessments will be conducted once)
  The 'Practitioner Competency Test' in the pre-test includes 5 questions
  Questions are:
  How confident are you in performing blood pressure measurements? How prepared do you feel for performing blood pressure measurements? How adequate is your practical knowledge for blood pressure measurements? How accurate do you think your blood pressure measurements are? How functional is the theoretical training received on blood pressure measurement during practice?
  These questions use a Visual Analog Scale for responses. Additionally, participants will answer statements about their confidence and knowledge in ECG skills using a 5-point Likert scale:
  "I feel confident in my ECG assessment skills." "I believe my practical knowledge for ECG application is sufficient." "I think I correctly assess ischemia and necrosis on an ECG." "I feel confident in ECG evaluation." "I find the theoretical training I received on ECG to be functional during practical application."
Theoretical Knowledge Level Assessment Test | One day (The assessments will be conducted once)
  The pre-test, prepared by the researchers and to be completed by all students before the simulation training, consists of a section called 'Theoretical Knowledge Level Assessment Test.' This section includes 3 open-ended questions designed to measure theoretical knowledge about blood pressure and ECG.
  The questions for blood pressure and ECG are as follows:
  What are the names of the first and last sounds heard during blood pressure measurement? What do these sounds signify? What are the normal blood pressure values in adults? Which artery is typically used for blood pressure measurement? What waves make up a normal ECG? What is the change seen on an ECG in myocardial ischemia? What are the changes seen on an ECG in myocardial infarction (necrosis)?

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided